CLINICAL TRIAL: NCT05786027
Title: Exploring the Feasibility of a Peer-Driven Intervention to Improve HIV Prevention Among Prisoners Who Inject Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000023524; 1K01DA047194-01 (NIH); 1K01DA047194-05 (NIH)
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: HIV

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Driven Intervention (PDI) (Experimental): Participants from two experimental (E) prisons that are HIV-negative will be assigned to this arm. Participants will receive 12 weeks of PDI and weekly opioid urine tests. Prior to intervention participants will receive training by a Health Educator (HE) in Health Advocate (HA) and Peer roles.
  Interventions: Behavioral: PDI
- Treatment As Usual (TAU) (No Intervention): Participants from two control (C) prisons that are HIV-negative will be assigned to this arm. Participants will receive treatment as usual (which includes universal access to SSP, MMT, and Atlantis program for individuals with opioid dependence) and weekly urine opioid tests for 12 weeks.

INTERVENTIONS:
Behavioral: PDI — A 12-week in-prison peer-driven intervention to increase the uptake of primary HIV prevention strategies (readiness to initiate addiction treatment (MMT or Atlantis), initiation of MMT/Atlantis, retention in MMT/Atlantis; or the use of SSP), and reduce the use of opioids and HIV risk behaviors, in HIV-negative PWID in prison.
  Arms: Peer Driven Intervention (PDI)

SUMMARY:
The purpose of this study is to develop, conduct, and assess the feasibility of a) a pilot peer-driven intervention (PDI) to reduce HIV risk and increase the uptake of primary HIV prevention services (i.e. prison addiction treatment programs), and b) explore the PDI's usefulness from the perspective of both prisoners and prison staff to make recommendations for the PDI future improvement and adaptation.

DETAILED DESCRIPTION:
The investigators will develop and pilot a 12-week in-prison peer-driven intervention to increase the uptake of primary HIV prevention strategies (readiness to initiate addiction treatment (MMT or Atlantis), initiation of MMT/Atlantis, retention in MMT/Atlantis; or the use of SSP), and reduce the use of opioids and HIV risk behaviors, in HIV-negative PWID in prison.

Aim 1: To develop, conduct, and assess the feasibility and the immediate and durable effects of a 12-week within-prison PDI to reduce HIV risk and increase uptake of primary HIV prevention among prisoners who abuse drugs and are ≥1 year prior to release at baseline. The quasi-experimental design where two prisons will be assigned to experiment and two comparable prisons will be assigned to control, will strive to account for the potential threats to internal validity (e.g. history and maturation), and to external validity (e.g. various interaction effects between characteristics of selected participants and their engagement in HIV prevention). The focus of this registration is Aim 1.

Aim 2: Using the data from structured ethnographic observation of PDI sessions, and qualitative interviews immediately after the PDI with prisoner participants, staff of prison addiction treatment programs, and researchers who implemented the PDI, to explore why the PDI is successful (or not), and optimize the PDI manual.

ELIGIBILITY:
Inclusion Criteria:

* HIV negative by self-report before the study confirmed by HIV rapid test
* Has ever injected drugs
* ≥1 year before prison release (release dates are fixed and accurate)
* currently not enrolled in MMT/Atlantis
* Capable of providing informed consent.

Exclusion Criteria:

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — There is only one female prison in KYR and few women PWID in prison (about 1% of the total female prisoner population) per our recent bio-behavioral study. Thus, only men will be included into the pilot PDI in this instance.
Enrollment: 100 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Number of participants enrolled in MMT or Atlantis 12-step addiction recovery program | up to 12 weeks
  Number of participants that enrolled in MMT or Atlantis 12-step addiction recovery program from baseline up to 12 weeks.
Number of participants enrolled in MMT or Atlantis 12-step addiction recovery program | Month 9
  Number of participants that enrolled in MMT or Atlantis 12-step addiction recovery program at month 9.

SECONDARY OUTCOMES:
Number of times participants relapsed | Month 6
  Number of times participants had any kind of relapse at Month 6.
Number of times participants relapsed | Month 9
  Number of times participants had any kind of relapse at Month 9.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Rozanova, PhD, Principal Investigator — Yale University
Locations (1):
- Prison System, Bishkek, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT05786027/ICF_000.pdf